CLINICAL TRIAL: NCT02714595
Title: A Multicenter, Randomized, Open-label Clinical Study of S-649266 or Best Available Therapy for the Treatment of Severe Infections Caused by Carbapenem-resistant Gram-negative Pathogens
Brief Title: Study of Cefiderocol (S-649266) or Best Available Therapy for the Treatment of Severe Infections Caused by Carbapenem-resistant Gram-negative Pathogens
Acronym: CREDIBLE - CR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1424R2131; 2015-004703-23 (EudraCT Number)
Expanded Access: NCT03780140 (Approved for marketing)
Record Dates: First submitted 2016-02-26; First posted 2016-03-21 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2020-12

CONDITIONS: Healthcare-associated Pneumonia (HCAP); Bloodstream Infections (BSI); Hospital Acquired Pneumonia (HAP); Complicated Urinary Tract Infection (cUTI); Sepsis; Ventilator Associated Pneumonia (VAP)
Keywords: cefiderocol; Bloodstream infections (BSI); Complicated urinary tract infection (cUTI); Ventilator associated pneumonia (VAP); Hospital acquired pneumonia (HAP); Sepsis; multi-drug resistant pathogens; S-649266; Gram-negative pathogens; Healthcare-associated pneumonia (HCAP); carbapenem resistant pathogens
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Sepsis; Pneumonia, Ventilator-Associated | interventions — Cefiderocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cefiderocol (Experimental): Participants will receive cefiderocol 2 g administered intravenously over 3 hours, every 8 hours for 7-14 days. Treatment could be extended to 21 days at the discretion of the investigator.
  Interventions: Drug: Cefiderocol
- Best Available Therapy (BAT) (Active Comparator): Best available therapy (BAT) will be chosen by the investigator and may include up to three antibacterial agents for carbapenem resistant Gram-negative bacteria, intravenously administered per country-specific guidelines for 7-14 days. Treatment could be extended to 21 days at the discretion of the investigator.
  Interventions: Drug: Best Available Therapy

INTERVENTIONS:
Drug: Cefiderocol — 2 g intravenously over 3 hours every 8 hours for a period of 7 to 14 days, or 2 g every 6 hours for participants with creatinine clearance >120 mL/min.
  Other Names: S-649266; Fetroja ®
  Arms: Cefiderocol
Drug: Best Available Therapy — Standard of care with either a polymyxin-based or non-polymyxin-based regimen as determined by the investigator and consisting of one to three marketed antibacterial agent(s).
  Arms: Best Available Therapy (BAT)

SUMMARY:
This study is designed to provide evidence of efficacy of cefiderocol in the treatment of serious infections in adult patients caused by carbapenem-resistant Gram-negative pathogens.

DETAILED DESCRIPTION:
This study is designed to provide evidence of efficacy of cefiderocol in the treatment of serious infections in adult patients with either hospital-acquired pneumonia (HAP), ventilator-associated pneumonia (VAP), healthcare-associated pneumonia (HCAP), complicated urinary tract infection (cUTI), or bloodstream infections (BSI)/sepsis caused by carbapenem-resistant Gram-negative pathogens.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically documented infection (HAP/VAP/HCAP, cUTI, or BSI/sepsis) caused by a Gram-negative pathogen with evidence of carbapenem resistance
* Patients who have been treated previously with an empiric antibiotic regiment and failed treatment, both clinically and microbiologically, are eligible for the study, if they have an identified carbapenem-resistant Gram-negative pathogen which has either been shown to be nonsusceptible in vitro to each of the antibiotic(s) of the empiric antibiotic regimen or been grown from a culture performed after at least 2 days of the empiric antibiotic regimen
* Patient is male (no contraception required) or female and meets one of the following criteria:

  * Surgically sterile by hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy or tubal ligation for the purpose of contraception for at least 6 weeks with appropriate documentation of such surgery
  * Postmenopausal (defined as older than 45 years of age with cessation of regular menstrual periods for 6 months and confirmed by a follicle-stimulating hormone level of > 40 mIU/mL, or amenorrhea for at least 12 months)
  * Of childbearing potential and using combined (estrogen and progestogen) or progestogen-only hormonal contraception associated with inhibition of ovulation (including oral, intravaginal, injectable, implantable, and transdermal contraceptives), or an intrauterine device (IUD), or intrauterine hormone-releasing system (IUS) for the entire duration of the study
  * Of childbearing potential and practice abstinence as a preferred and usual lifestyle, and agrees to continue practicing abstinence from Screening and for the entire duration of the study
  * Of childbearing potential, whose sole heterosexual partner has been successfully vasectomized and agrees to not have other heterosexual partners for the entire duration of the study
* Patients meeting specific criteria for each infection site

Exclusion Criteria:

1. Patients who have a history of any moderate or severe hypersensitivity or allergic reaction to any β-lactam (Note: for β-lactams, a history of a mild rash followed by uneventful re-exposure is not a contraindication to enrollment)
2. Patients who need more than 3 systemic antibiotics as part of best available therapy (BAT) for the treatment of the Gram-negative infection (patients with mixed Gram-positive or anaerobic infections may receive appropriate concomitant narrow spectrum antibiotics [eg, vancomycin, linezolid, metronidazole, clindamycin])
3. Patients with coinfection caused by invasive aspergillosis, mucormycosis or other highly lethal mold
4. Patients who have central nervous system (CNS) infection (eg, meningitis, brain abscess, shunt infection)
5. Patients with infection requiring > 3 weeks of antibiotic treatment (eg, bone and joint infection, endocarditis)
6. Patients with cystic fibrosis or moderate to severe bronchiectasis
7. Patients in refractory septic shock defined as persistent hypotension despite adequate fluid resuscitation or despite vasopressive therapy at the time of Randomization
8. Patients with severe neutropenia, ie, polymorphonuclear neutrophils (PMNs) < 100 cells/μL
9. Female patients who have a positive pregnancy test at Screening or who are lactating
10. Patients with Acute Physiology and Chronic Health Evaluation II (APACHE II) score > 30
11. Patients who have received a potentially effective antibiotic regimen for the carbapenem-resistant Gram-negative infection for a continuous duration of more than 24 hours in cUTI, or 36 hours in HAP/VAP/HCAP or BSI/sepsis during the 72 hours leading to Randomization
12. Patients with any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the patient or the quality of the study data
13. Patients who have received another investigational drug or device within 30 days prior to study entry
14. Patients who have previously been randomized in this study or received S-649266
15. Patients receiving peritoneal dialysis
16. Patients meeting specific exclusion criteria for each infection site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shionogi Clinical Trials Administrator Clinical Support Help Line, Study Director — Shionogi
Locations (69):
- United States (6):
  - Shionogi Research Site, Hartford, Connecticut
  - Shionogi Research Site, Newark, Delaware
  - Shionogi Research Site, Chicago, Illinois
  - Shionogi Research Site, New Orleans, Louisiana
  - Shionogi Research Site, Detroit, Michigan
  - Shionogi Research Site, Pittsburgh, Pennsylvania
- Brazil (7):
  - Shionogi Research Site, Salvador, Estado de Bahia
  - Shionogi Research Site, Curitiba, Paraná
  - Shionogi Research Site, Passo Fundo, Rio Grande do Sul
  - Shionogi Research Site, Porto Alegre, Rio Grande do Sul
  - Shionogi Research Site, Santa Maria, Rio Grande do Sul
  - Shionogi Research Site, São José do Rio Preto, São Paulo
  - Shionogi Research Site, São Paulo, São Paulo
- Croatia (3):
  - Shionogi Research Site, Rijeka, Primorje-Gorski Kotar County
  - Shionogi Research Site, Split
  - Shionogi Research Site, Zagreb
- France (2):
  - Shionogi Research Site, La Tronche, Auvergne-Rhône-Alpes
  - Shionogi Research Site, Paris, Île-de-France Region
- Germany (3):
  - Shionogi Research Site, Heidelberg, Baden-Wurttemberg
  - Shionogi Research Site, Bonn, North Rhine-Westphalia
  - Shionogi Research Site, Berlin
- Greece (3):
  - Shionogi Research Site, Athens, Attica
  - Shionogi Research Site, Patra, Peloponnese
  - Shionogi Research Site, Larissa, Thessaly
- Shionogi Research Site, Guatemala City, Guatemala
- Israel (9):
  - Shionogi Research Site, Beersheba, Beersheba
  - Shionogi Research Site, Be’er Ya‘aqov, Rehoboth
  - Shionogi Research Site, Tel Aviv, Tel Aviv
  - Shionogi Research Site, Tel Litwinsky, Tel Aviv
  - Shionogi Research Site, Safed, Zefat
  - Shionogi Research Site, Hadera
  - Shionogi Research Site, Haifa
  - Shionogi Research Site, Holon
  - Shionogi Research Site, Jerusalem
- Italy (4):
  - Shionogi Research Site, Cisanello, PISA
  - Shionogi Research Site, Milan
  - Shionogi Research Site, Modena
  - Shionogi Research Site, Udine
- Japan (3):
  - Shionogi Research Site, Nagakute, Aichi-ken
  - Shionogi Research Site, Shinagawa-ku, Tokyo
  - Shionogi Research Site, Nagasaki
- South Korea (4):
  - Shionogi Research Site, Wŏnju, Gangwon-do
  - Shionogi Research Site, Seoul, Gwangjin-gu
  - Shionogi Research Site, Daegu
  - Shionogi Research Site, Seoul
- Spain (11):
  - Shionogi Research Site, Terrassa, Barcelona
  - Shionogi Research Site, Córdoba, Cordoba
  - Shionogi Research Site, Lleida, Lleida
  - Shionogi Research Site, Barcelona
  - Shionogi Research Site, Ciudad Real
  - Shionogi Research Site, Girona
  - Shionogi Research Site, Madrid
  - Shionogi Research Site, Málaga
  - Shionogi Research Site, Seville
  - Shionogi Research Site, Valencia
  - Shionogi Research Site, Zaragoza
- Taiwan (5):
  - Shionogi Research Site, Hualien City, Hualien
  - Shionogi Research Site, Taichung, ROC
  - Shionogi Research Site, Taipei City, Taipei
  - Shionogi Research Site, Kaohsiung City
  - Shionogi Research Site, Taichung
- Thailand (3):
  - Shionogi Research Site, Bangkok
  - Shionogi Research Site, Muang Nonthaburi
  - Shionogi Research Site, Muang
- Turkey (Türkiye) (4):
  - Shionogi Research Site, Bornova, İzmir
  - Shionogi Research Site, Ankara
  - Shionogi Research Site, Istanbul
  - Shionogi Research Site, Trabzon
- Shionogi Research Site, London, England, United Kingdom

REFERENCES:
- [Derived] Nordmann P, Shields RK, Doi Y, Takemura M, Echols R, Matsunaga Y, Yamano Y. Mechanisms of Reduced Susceptibility to Cefiderocol Among Isolates from the CREDIBLE-CR and APEKS-NP Clinical Trials. Microb Drug Resist. 2022 Apr;28(4):398-407. doi: 10.1089/mdr.2021.0180. Epub 2022 Jan 24. PMID 35076335
- [Derived] Wenzler E, Butler D, Tan X, Katsube T, Wajima T. Pharmacokinetics, Pharmacodynamics, and Dose Optimization of Cefiderocol during Continuous Renal Replacement Therapy. Clin Pharmacokinet. 2022 Apr;61(4):539-552. doi: 10.1007/s40262-021-01086-y. Epub 2021 Nov 18. PMID 34792787
- [Derived] Naseer S, Weinstein EA, Rubin DB, Suvarna K, Wei X, Higgins K, Goodwin A, Jang SH, Iarikov D, Farley J, Nambiar S. US Food and Drug Administration (FDA): Benefit-Risk Considerations for Cefiderocol (Fetroja(R)). Clin Infect Dis. 2021 Jun 15;72(12):e1103-e1111. doi: 10.1093/cid/ciaa1799. PMID 33393598
- [Derived] Bassetti M, Echols R, Matsunaga Y, Ariyasu M, Doi Y, Ferrer R, Lodise TP, Naas T, Niki Y, Paterson DL, Portsmouth S, Torre-Cisneros J, Toyoizumi K, Wunderink RG, Nagata TD. Efficacy and safety of cefiderocol or best available therapy for the treatment of serious infections caused by carbapenem-resistant Gram-negative bacteria (CREDIBLE-CR): a randomised, open-label, multicentre, pathogen-focused, descriptive, phase 3 trial. Lancet Infect Dis. 2021 Feb;21(2):226-240. doi: 10.1016/S1473-3099(20)30796-9. Epub 2020 Oct 12. PMID 33058795
- [Derived] Bassetti M, Ariyasu M, Binkowitz B, Nagata TD, Echols RM, Matsunaga Y, Toyoizumi K, Doi Y. Designing A Pathogen-Focused Study To Address The High Unmet Medical Need Represented By Carbapenem-Resistant Gram-Negative Pathogens - The International, Multicenter, Randomized, Open-Label, Phase 3 CREDIBLE-CR Study. Infect Drug Resist. 2019 Nov 21;12:3607-3623. doi: 10.2147/IDR.S225553. eCollection 2019. PMID 31819544

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled hospitalized patients with hospital-acquired pneumonia (HAP), ventilator-associated pneumonia (VAP), healthcare-associated pneumonia (HCAP), bloodstream infection (BSI), sepsis, or complicated urinary tract infection (cUTI) caused by carbapenem-resistant Gram-negative pathogens, and was conducted at 95 sites in 16 countries.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive therapy with cefiderocol or best available therapy (BAT), stratified by primary clinical diagnosis (HAP/VAP/HCAP, BSI/sepsis, cUTI), Acute Physiology and Chronic Health Evaluation (APACHE) II score (≤ 15 or ≥ 16-≤ 30), and region (North America, South America region, Europe, Asia-Pacific).
Groups:
- Cefiderocol: Participants received 2 g cefiderocol administered intravenously over 3 hours, every 8 hours for 7-14 days.
- Best Available Therapy (BAT): Participants received best available therapy, as chosen by the investigator, and may have included up to three antibacterial agents for carbapenem resistant Gram-negative bacteria, intravenously administered per country-specific guidelines for 7-14 days.
Period: Overall Study
Arm/Group | Cefiderocol | Best Available Therapy (BAT)
Started | 101 | 51
Received Treatment (Safety population) | 101 | 49
Carbapenem-resistant Microbiological Intent-to-treat (CR Micro-ITT population; See definition in Baseline Characteristics section) | 80 | 38
Completed | 69 | 38
Not Completed | 32 | 13
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Death | 30 | 9
Not completed — Other-Miscellaneous | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Carbapenem-resistant Microbiological Intent-to-treat (CR Micro-ITT) population includes randomized participants who received at least 1 dose of study drug and who had a central laboratory confirmed carbapenem resistant Gram-negative pathogen at Baseline from an appropriate clinical biospecimen.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefiderocol | Best Available Therapy (BAT) | Total
Number analyzed (Participants) | 80 | 38 | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (18.7) | 62.1 (17.3) | 62.8 (18.2)
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 30 | 21 | 51
  ≥ 65 years | 50 | 17 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 9 | 34
  Male | 55 | 29 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 2 | 12
  Not Hispanic or Latino | 64 | 35 | 99
  Unknown or Not Reported | 6 | 1 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 48 | 27 | 75
  Asian | 24 | 9 | 33
  Other | 8 | 2 | 10
Region [Count of Participants; unit: Participants]
  North America | 4 | 3 | 7
  South America | 7 | 3 | 10
  Europe | 45 | 23 | 68
  Asia-Pacific | 24 | 9 | 33
Total APACHE II Score [Count of Participants; unit: Participants] — Acute Physiology And Chronic Health Evaluation II is a severity-of-disease classification applied within 24 hours of admission of a patient to an intensive care unit (ICU). The APACHE II score consists of three parts: 12 acute physiological variables, age, and chronic health status. The range of the score is 0 to 71, where higher scores correspond to more severe disease and a higher risk of death.
  Participants
    ≤ 15 | 41 | 21 | 62
    ≥ 16 | 39 | 17 | 56
Clinical Diagnosis [Count of Participants; unit: Participants] — BSI = bloodstream infection; cUTI = complicated urinary tract infection; HAP = hospital-acquired pneumonia; HCAP = healthcare-associated pneumonia; VAP = ventilator-associated pneumonia
  Participants
    HAP/VAP/HCAP | 40 | 19 | 59
    BSI/Sepsis | 23 | 14 | 37
    cUTI | 17 | 5 | 22
Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: units on a scale] — The SOFA score is a scoring system to determine the extent of a patient's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems. Each score is from 0 to 4, the total score ranges from 0 to 24, where higher scores indicate a higher likelihood of mortality.
  units on a scale | 5.6 (4.1) | 5.6 (3.9) | 5.6 (4.0)
Clinical Pulmonary Infection Score (CPIS) [Mean (Standard Deviation); unit: units on a scale] — Clinical pulmonary infection score (CPIS) is a surrogate for diagnosis and treatment response. Points (0, 1, or 2) are assigned for observed findings for 5 variables including body temperature, white blood cell count, tracheal secretions, ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2) and chest radiograph infiltrates.
  The total score ranges from 0 to 10, where higher scores may indicate a higher likelihood of mortality. Population: Only conducted in participants with HAP/VAP/HCAP; 2 participants had missing CPIS scores at Baseline.
  units on a scale
    number analyzed (Participants) | 39 | 18 | 57
    (all) | 5.1 (1.6) | 5.0 (1.1) | 5.1 (1.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Cure at Test of Cure (TOC) in Participants With HAP/VAP/HCAP or BSI/Sepsis
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms and was defined for each diagnosis.
  HAP/VAP/HCAP: Clinical cure was defined as resolution or substantial improvement of Baseline signs and symptoms of pneumonia including a reduction in SOFA and CPIS scores, and improvement or lack of progression of chest radiographic abnormalities such that no antibacterial therapy was required for the treatment of the current infection.
  BSI/Sepsis: Clinical cure was defined as resolution or substantial improvement of Baseline signs and symptoms including a reduction in SOFA score, such that no antibacterial therapy was required for the treatment of BSI/sepsis. Participants with bacteremia must have eradication of bacteremia caused by the Gram-negative pathogen.
  Participants with missing data were considered as non-responders.
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: Carbapenem-resistant Microbiological Intent-to-treat (CR Micro-ITT) Population included all participants who received at least 1 dose of the study treatment, who had a baseline Gram-negative pathogen from an appropriate clinical specimen, and whose baseline Gram-negative pathogen was carbapenem-resistant as confirmed by central laboratory testing.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HAP/VAP/HCAP: Cefiderocol: Participants with HAP/VAP/HCAP received 2 g cefiderocol administered intravenously over 3 hours, every 8 hours for 7-14 days.
- HAP/VAP/HCAP: Best Available Therapy: Participants with HAP/VAP/HCAP received best available therapy, as chosen by the investigator, which may have included up to three antibacterial agents for carbapenem resistant Gram-negative bacteria, intravenously administered per country-specific guidelines for 7-14 days.
- BSI/Sepsis: Cefiderocol: Participants with BSI/sepsis received 2 g cefiderocol administered intravenously over 3 hours, every 8 hours for 7-14 days.
- BSI/Sepsis: Best Available Therapy: Participants with BSI/sepsis received best available therapy, as chosen by the investigator, which may have included up to three antibacterial agents for carbapenem resistant Gram-negative bacteria, intravenously administered per country-specific guidelines for 7-14 days.
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14
percentage of participants | 50.0 [33.8 to 66.2] | 52.6 [28.9 to 75.6] | 43.5 [23.2 to 65.5] | 42.9 [17.7 to 71.1]

2. Primary Outcome: Percentage of Participants With Microbiologic Eradication at TOC in Participants With cUTI
Description: Microbiological outcome per Baseline pathogen was determined by the sponsor as defined for each infection site. For cUTI eradication was defined as a urine culture that showed that the Gram-negative uropathogen identified at Baseline at ≥ 10⁵ colony-forming units (CFU)/mL was reduced to < 10³ CFU/mL.
  Overall per-participant eradication was defined as eradication of all Baseline Gram-negative pathogens.
Time Frame: Test of cure, defined as 7 days after the end of treatment, equivalent to Study Days 14 to 21
Population: Carbapenem-resistant Microbiological Intent-to-treat Population; participants with missing data were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- cUTI: Cefiderocol: Participants with cUTI received 2 g cefiderocol administered intravenously over 3 hours, every 8 hours for 7-14 days.
- cUTI: Best Available Therapy: Participants with cUTI received best available therapy, as chosen by the investigator, and may have included up to three antibacterial agents for carbapenem resistant Gram-negative bacteria, intravenously administered per country-specific guidelines for 7-14 days.
Arm/Group | cUTI: Cefiderocol | cUTI: Best Available Therapy
Number analyzed (Participants) | 17 | 5
percentage of participants | 52.9 [27.8 to 77.0] | 20.0 [0.5 to 71.6]

3. Secondary Outcome: Percentage of Participants With Clinical Cure at End of Treatment (EOT) in Participants With HAP/VAP/HCAP or BSI/Sepsis
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms and was defined for each diagnosis.
  HAP/VAP/HCAP: Clinical cure was defined as resolution or substantial improvement of Baseline signs and symptoms of pneumonia including a reduction in SOFA and CPIS scores, and improvement or lack of progression of chest radiographic abnormalities such that no antibacterial therapy was required for the treatment of the current infection.
  BSI/Sepsis: Clinical cure was defined as resolution or substantial improvement of Baseline signs and symptoms including a reduction in SOFA score, such that no antibacterial therapy was required for the treatment of BSI/sepsis. Participants with bacteremia must have eradication of bacteremia caused by the Gram-negative pathogen.
Time Frame: End of treatment, Day 7 to 14
Population: Carbapenem-resistant Microbiological Intent-to-treat Population; participants with missing data were counted as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14
percentage of participants | 60.0 [43.3 to 75.1] | 63.2 [38.4 to 83.7] | 69.6 [47.1 to 86.8] | 50.0 [23.0 to 77.0]

4. Secondary Outcome: Percentage of Participants With Sustained Clinical Cure at Follow-up (FU) in Participants With HAP/VAP/HCAP or BSI/Sepsis
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms and was defined for each diagnosis.
  Sustained clinical cure for HAP/VAP/HCAP: Continued resolution or substantial improvement of Baseline signs and symptoms of pneumonia, such that no antibacterial therapy was required for the treatment of pneumonia in a participant assessed as cured at TOC.
  BSI/Sepsis: Continued resolution or substantial improvement of Baseline signs and symptoms associated with reduction in SOFA score, such that no antibacterial therapy was required for the treatment of the original BSI/sepsis in a participant assessed as cured at TOC.
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14
percentage of participants | 50.0 [33.8 to 66.2] | 31.6 [12.6 to 56.6] | 39.1 [19.7 to 61.5] | 28.6 [8.4 to 58.1]

5. Secondary Outcome: Percentage of Participants With Clinical Cure at Test of Cure in Participants With cUTI
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms and was defined for each diagnosis.
  cUTI: Resolution or substantial improvement of Baseline signs and symptoms of cUTI, or return to pre-infection Baseline if known, such that no antibacterial therapy is required for the treatment of the current infection.
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | cUTI: Cefiderocol | cUTI: Best Available Therapy
Number analyzed (Participants) | 17 | 5
percentage of participants | 70.6 [44.0 to 89.7] | 60.0 [14.7 to 94.7]

6. Secondary Outcome: Percentage of Participants With Clinical Cure at End of Treatment (EOT) in Participants With cUTI
Description: as for outcome 5
Time Frame: End of treatment, Day 7 to 14
Population: Carbapenem-resistant Microbiological Intent-to-treat Population; participants with missing data were considered as non-responders
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | cUTI: Cefiderocol | cUTI: Best Available Therapy
Number analyzed (Participants) | 17 | 5
percentage of participants | 76.5 [50.1 to 93.2] | 60.0 [14.7 to 94.7]

7. Secondary Outcome: Percentage of Participants With Sustained Clinical Cure at Follow-up in Participants With cUTI
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms and was defined for each diagnosis.
  Sustained clinical cure for cUTI: Continued resolution or improvement of Baseline signs and symptoms of cUTI, or return to pre-infection Baseline if known, in a participant assessed as cured at TOC.
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: Carbapenem-resistant Microbiological Intent-to-treat Population); participants with missing data were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | cUTI: Cefiderocol | cUTI: Best Available Therapy
Number analyzed (Participants) | 17 | 5
percentage of participants | 52.9 [27.8 to 77.0] | 60.0 [14.7 to 94.7]

8. Secondary Outcome: Percentage of Participants With Clinical Cure at End of Treatment in Participants With HAP/VAP/HCAP + BSI/Sepsis, and Overall
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms and was defined for each diagnosis.
  HAP/VAP/HCAP: Resolution or substantial improvement of Baseline signs and symptoms of pneumonia including a reduction in SOFA and CPIS scores, and improvement or lack of progression of chest radiographic abnormalities such that no antibacterial therapy was required for the treatment of the current infection.
  BSI/Sepsis: Resolution or substantial improvement of Baseline signs and symptoms including a reduction in SOFA score, such that no antibacterial therapy was required for the treatment of BSI/sepsis. Participants with bacteremia must have eradication of bacteremia caused by the Gram-negative pathogen.
  cUTI: Resolution or substantial improvement of Baseline signs and symptoms of cUTI, or return to pre-infection Baseline if known, such that no antibacterial therapy is required for the treatment of the current infection.
Time Frame: End of treatment, Day 7 to 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol: Participants with HAP/VAP/HCAP or BSI/sepsis received 2 g cefiderocol administered intravenously over 3 hours, every 8 hours for 7-14 days.
- HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy: Participants with HAP/VAP/HCAP or BSI/sepsis received best available therapy, as chosen by the investigator, which may have included up to three antibacterial agents for carbapenem resistant Gram-negative bacteria, intravenously administered per country-specific guidelines for 7-14 days.
- Overall: Cefiderocol: Participants with HAP/VAP/HCAP, BSI/sepsis, or cUTI received 2 g cefiderocol administered intravenously over 3 hours, every 8 hours for 7-14 days.
- Overall: Best Available Therapy: Participants with HAP/VAP/HCAP, BSI/sepsis, or cUTI received best available therapy, as chosen by the investigator, which may have included up to three antibacterial agents for carbapenem resistant Gram-negative bacteria, intravenously administered per country-specific guidelines for 7-14 days.
Arm/Group | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 63 | 33 | 80 | 38
percentage of participants | 63.5 [50.4 to 75.3] | 57.6 [39.2 to 74.5] | 66.3 [54.8 to 76.4] | 57.9 [40.8 to 73.7]

9. Secondary Outcome: Percentage of Participants With Clinical Cure at Test of Cure in Participants With HAP/VAP/HCAP + BSI/Sepsis, and Overall
Description: as for outcome 8
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 63 | 33 | 80 | 38
percentage of participants | 47.6 [34.9 to 60.6] | 48.5 [30.8 to 66.5] | 52.5 [41.0 to 63.8] | 50.0 [33.4 to 66.6]

10. Secondary Outcome: Percentage of Participants With Sustained Clinical Cure at Follow-up in Participants With HAP/VAP/HCAP + BSI/Sepsis, and Overall
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms and was defined for each diagnosis.
  Sustained clinical cure for HAP/VAP/HCAP: Continued resolution or substantial improvement of Baseline signs and symptoms of pneumonia, such that no antibacterial therapy is required for the treatment of pneumonia in a participant assessed as cured at TOC.
  BSI/Sepsis: Continued resolution or substantial improvement of Baseline signs and symptoms associated with reduction in SOFA score, such that no antibacterial therapy is required for the treatment of the original BSI/sepsis in a participant assessed as cured at TOC.
  cUTI: Continued resolution or improvement of Baseline signs and symptoms of cUTI, or return to pre-infection Baseline if known, in a participant assessed as cured at TOC.
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 63 | 33 | 80 | 38
percentage of participants | 46.0 [33.4 to 59.1] | 30.3 [15.6 to 48.7] | 47.5 [36.2 to 59.0] | 34.2 [19.6 to 51.4]

11. Secondary Outcome: Percentage of Participants With Clinical Cure at End of Treatment By Baseline Pathogen
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms and was defined for each diagnosis:
  HAP/VAP/HCAP: Resolution or substantial improvement of Baseline signs and symptoms of pneumonia including a reduction in SOFA and CPIS scores, and improvement or lack of progression of chest radiographic abnormalities such that no antibacterial therapy was required for the treatment of the current infection.
  BSI/Sepsis: Resolution or substantial improvement of Baseline signs and symptoms including a reduction in SOFA score, such that no antibacterial therapy was required for the treatment of BSI/sepsis. Participants with bacteremia must have eradication of bacteremia caused by the Gram-negative pathogen.
  cUTI: Resolution or substantial improvement of Baseline signs and symptoms of cUTI, or return to pre-infection Baseline if known, such that no antibacterial therapy is required for the treatment of the current infection.
Time Frame: End of treatment, Day 7 to 14
Population: Carbapenem-resistant Microbiological Intent-to-treat Population with the relevant pathogen at Baseline; participants with missing data were considered non-responders.
Measure: Number; unit: percentage of participants
Groups:
- cUTI: Best Available Therapy: Participants with cUTI received best available therapy, as chosen by the investigator, which may have included up to three antibacterial agents for carbapenem resistant Gram-negative bacteria, intravenously administered per country-specific guidelines for 7-14 days.
- Overall: Cefiderocol: Participants received 2 g cefiderocol administered intravenously over 3 hours, every 8 hours for 7-14 days.
- Overall: Best Available Therapy: Participants received best available therapy, as chosen by the investigator, which may have included up to three antibacterial agents for carbapenem resistant Gram-negative bacteria, intravenously administered per country-specific guidelines for 7-14 days.
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 61.5 | 70.0 | 70.0 | 42.9 | 0 |  | 63.9 | 58.8 | 62.2 | 58.8
  Pseudomonas aeruginosa: number analyzed (Participants) | 11 | 6 | 2 | 3 | 4 | 2 | 13 | 9 | 17 | 11
  Pseudomonas aeruginosa | 63.6 | 83.3 | 100.0 | 33.3 | 50.0 | 50.0 | 69.2 | 66.7 | 64.7 | 63.6
  Klebsiella pneumoniae: number analyzed (Participants) | 10 | 5 | 11 | 4 | 11 | 3 | 21 | 9 | 32 | 12
  Klebsiella pneumoniae | 70.0 | 40.0 | 63.6 | 75.0 | 90.9 | 66.7 | 66.7 | 55.6 | 75.0 | 58.3
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 20.0 |  |  |  |  |  | 20.0 |  | 20.0 |
  Escherichia coli: number analyzed (Participants) | 2 | 2 | 2 | 0 | 1 | 0 | 4 | 2 | 5 | 2
  Escherichia coli | 100.0 | 0 | 100.0 |  | 100.0 |  | 100.0 | 0 | 100.0 | 0

12. Secondary Outcome: Percentage of Participants With Clinical Cure at Test of Cure By Baseline Pathogen
Description: as for outcome 8
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 50.0 | 60.0 | 30.0 | 42.9 | 0 |  | 44.4 | 52.9 | 43.2 | 52.9
  Pseudomonas aeruginosa: number analyzed (Participants) | 11 | 6 | 2 | 3 | 4 | 2 | 13 | 9 | 17 | 11
  Pseudomonas aeruginosa | 45.5 | 66.7 | 100.0 | 33.3 | 50.0 | 50.0 | 53.8 | 55.6 | 52.9 | 54.5
  Klebsiella pneumoniae: number analyzed (Participants) | 10 | 5 | 11 | 4 | 11 | 3 | 21 | 9 | 32 | 12
  Klebsiella pneumoniae | 60.0 | 40.0 | 54.5 | 50.0 | 81.8 | 66.7 | 57.1 | 44.4 | 65.6 | 50.0
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 0.0 |  |  |  |  |  | 5.0 |  | 0.0 |
  Escherichia coli: number analyzed (Participants) | 2 | 2 | 2 | 0 | 1 | 0 | 4 | 2 | 5 | 2
  Escherichia coli | 50.0 | 0.0 | 50.0 |  | 100.0 |  | 50.0 | 0.0 | 60.0 | 0.0

13. Secondary Outcome: Percentage of Participants With Sustained Clinical Cure at Follow-up By Baseline Pathogen
Description: Clinical response was based on the investigator's evaluation of the participant's clinical signs and symptoms and was defined for each diagnosis.
  Sustained clinical cure for HAP/VAP/HCAP: Continued resolution or substantial improvement of Baseline signs and symptoms of pneumonia, such that no antibacterial therapy was required for the treatment of pneumonia in a participant assessed as cured at TOC.
  BSI/Sepsis: Continued resolution or substantial improvement of Baseline signs and symptoms associated with reduction in SOFA score, such that no antibacterial therapy was required for the treatment of the original BSI/sepsis in a participant assessed as cured at TOC.
  cUTI: Continued resolution or improvement of Baseline signs and symptoms of cUTI, or return to pre-infection Baseline if known, in a participant assessed as cured at TOC.
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 50.0 | 60.0 | 30.0 | 28.6 | 0.0 |  | 44.4 | 35.3 | 43.2 | 35.3
  Pseudomonas aeruginosa: number analyzed (Participants) | 11 | 6 | 2 | 3 | 4 | 2 | 13 | 9 | 17 | 11
  Pseudomonas aeruginosa | 45.5 | 16.7 | 100.0 | 33.3 | 25.0 | 50.0 | 53.8 | 55.6 | 47.1 | 27.3
  Klebsiella pneumoniae: number analyzed (Participants) | 10 | 5 | 11 | 4 | 11 | 3 | 21 | 9 | 32 | 12
  Klebsiella pneumoniae | 60.0 | 40.0 | 45.5 | 25.0 | 63.6 | 66.7 | 52.4 | 33.3 | 56.3 | 41.7
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 0.0 |  |  |  |  |  | 0.0 |  | 0.0 |
  Escherichia coli: number analyzed (Participants) | 2 | 2 | 2 | 0 | 1 | 0 | 4 | 2 | 5 | 2
  Escherichia coli | 50.0 | 0.0 | 50.0 |  | 100.0 |  | 50.0 | 0.0 | 60.0 | 0.0

14. Secondary Outcome: Percentage of Participants With Clinical Cure at EOT By Baseline Carbapenem-resistant Pathogen
Description: as for outcome 11
Time Frame: End of treatment, Day 7 to 14
Population: Carbapenem-resistant Microbiological Intent-to-treat Population with the relevant carbapenem-resistant pathogen at Baseline; participants with missing data were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 61.5 | 70.0 | 70.0 | 42.9 | 0.0 |  | 63.9 | 58.8 | 62.2 | 58.8
  Klebsiella pneumoniae: number analyzed (Participants) | 6 | 5 | 10 | 4 | 11 | 3 | 16 | 9 | 27 | 12
  Klebsiella pneumoniae | 83.3 | 40.0 | 60.0 | 75.0 | 90.9 | 66.7 | 68.8 | 55.6 | 77.8 | 58.3
  Pseudomonas aeruginosa: number analyzed (Participants) | 6 | 5 | 2 | 3 | 4 | 2 | 8 | 8 | 12 | 10
  Pseudomonas aeruginosa | 50.0 | 80.0 | 100.0 | 33.3 | 50.0 | 50.0 | 62.5 | 62.5 | 58.3 | 60.0
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 20.0 |  |  |  |  |  | 20.0 |  | 20.0 |

15. Secondary Outcome: Percentage of Participants With Clinical Cure at TOC By Baseline Carbapenem-resistant Pathogen
Description: as for outcome 11
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 50.0 | 60.0 | 30.0 | 42.9 | 0.0 |  | 44.4 | 52.9 | 43.2 | 52.9
  Klebsiella pneumoniae: number analyzed (Participants) | 6 | 5 | 10 | 4 | 11 | 3 | 16 | 9 | 27 | 12
  Klebsiella pneumoniae | 66.7 | 40.0 | 50.0 | 50.0 | 81.8 | 66.7 | 56.3 | 44.4 | 66.7 | 50.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 6 | 5 | 2 | 3 | 4 | 2 | 8 | 8 | 12 | 10
  Pseudomonas aeruginosa | 50.0 | 60.0 | 100.0 | 33.3 | 50.0 | 50.0 | 62.5 | 50.0 | 58.3 | 50.0
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 0.0 |  |  |  |  |  | 0.0 |  | 0.0 |

16. Secondary Outcome: Percentage of Participants With Sustained Clinical Cure at Follow-up By Baseline Carbapenem-resistant Pathogen
Description: as for outcome 13
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 50.0 | 40.0 | 30.0 | 28.6 | 0.0 |  | 44.4 | 35.3 | 43.2 | 35.3
  Klebsiella pneumoniae: number analyzed (Participants) | 6 | 5 | 10 | 4 | 11 | 3 | 16 | 9 | 27 | 12
  Klebsiella pneumoniae | 66.7 | 40.0 | 40.0 | 25.0 | 63.6 | 66.7 | 50.0 | 33.3 | 55.6 | 41.7
  Pseudomonas aeruginosa: number analyzed (Participants) | 6 | 5 | 2 | 3 | 4 | 2 | 8 | 8 | 12 | 10
  Pseudomonas aeruginosa | 50.0 | 20.0 | 100.0 | 33.3 | 25.0 | 50.0 | 62.5 | 25.0 | 50.0 | 30.0
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 0.0 |  |  |  |  |  | 0.0 |  | 0.0 |

17. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at EOT in Participants With HAP/VAP/HCAP or BSI/Sepsis
Description: Microbiological outcomes per Baseline pathogen were determined by the sponsor according to the following criteria established for each infection site:
  HAP/VAP/HCAP: Eradication was defined as the absence of the Baseline Gram-negative pathogen from an appropriate clinical specimen (sputum, tracheal aspirate, bronchoalveolar lavage (BAL) fluid, protected specimen brush, pleural fluid, or lung biopsy). If it was not possible to obtain an appropriate clinical culture and the participant had a successful clinical outcome, the response was presumed to be eradication.
  BSI/Sepsis: Absence of the Baseline Gram-negative pathogen from a blood culture and/or other primary source as applicable. In the case of sepsis, if the participant had a successful clinical outcome and it was not possible to obtain an appropriate clinical culture, the response was presumed to be eradication.
  Overall per-participant eradication was defined as eradication of all Baseline Gram-negative pathogens.
Time Frame: End of treatment, Day 7 to 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14
percentage of participants | 30.0 [16.6 to 46.5] | 26.3 [9.1 to 51.2] | 60.9 [38.5 to 80.3] | 28.6 [8.4 to 58.1]

18. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at TOC in Participants With HAP/VAP/HCAP or BSI/Sepsis
Description: as for outcome 17
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14
percentage of participants | 22.5 [10.8 to 38.5] | 21.1 [6.1 to 45.6] | 30.4 [13.2 to 52.9] | 28.6 [8.4 to 58.1]

19. Secondary Outcome: Percentage of Participants With Sustained Microbiologic Eradication at Follow-up in Participants With HAP/VAP/HCAP or BSI/Sepsis
Description: Microbiological outcomes per Baseline pathogen at FU were determined according to the following criteria for each diagnosis:
  HAP/VAP/HCAP: Sustained eradication was defined as the absence of the Baseline Gram-negative pathogen from an appropriate clinical specimen after TOC. If an appropriate clinical culture could not be obtained and the participant had a successful clinical response after TOC, the response was presumed sustained eradication.
  BSI/Sepsis: Absence of the Baseline Gram-negative pathogen from a blood culture or other primary source after TOC as applicable. For sepsis, if the participant has a successful clinical outcome after TOC and an appropriate clinical culture could not be obtained, the response was presumed sustained eradication.
  Overall per-participant response was defined as sustained eradication of all Baseline Gram-negative pathogens after documented eradication at TOC.
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14
percentage of participants | 20.0 [9.1 to 35.6] | 15.8 [3.4 to 39.6] | 26.1 [10.2 to 48.4] | 21.4 [4.7 to 50.8]

20. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at EOT in Participants With cUTI
Description: Microbiological outcome per Baseline pathogen was determined by the sponsor as defined for each infection site. For cUTI eradication was defined as a urine culture that showed that the Gram-negative uropathogen identified at Baseline at ≥ 10⁵ CFU/mL was reduced to < 10³ CFU/mL.
  Overall per-participant eradication was defined as eradication of all Baseline Gram-negative pathogens.
Time Frame: End of treatment, Day 7 to 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | cUTI: Cefiderocol | cUTI: Best Available Therapy
Number analyzed (Participants) | 17 | 5
percentage of participants | 70.6 [44.0 to 89.7] | 20.0 [0.5 to 71.6]

21. Secondary Outcome: Percentage of Participants With Sustained Microbiologic Eradication at Follow-up in Participants With cUTI
Description: Microbiological outcome per Baseline pathogen at follow-up was determined by the sponsor as defined for each infection site.
  For cUTI sustained eradication was defined as a culture taken any time after documented eradication at TOC and a urine culture obtained at FU showed that the Baseline uropathogen found at entry at ≥10⁵ CFU/mL remained <10³ CFU/mL.
  Overall per-participant sustained eradication was defined as sustained eradication of all Baseline Gram-negative pathogens.
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | cUTI: Cefiderocol | cUTI: Best Available Therapy
Number analyzed (Participants) | 17 | 5
percentage of participants | 41.2 [18.4 to 67.1] | 20.0 [0.5 to 71.6]

22. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at EOT in Participants With HAP/VAP/HCAP + BSI/Sepsis, and Overall
Description: Microbiological outcomes per Baseline pathogen were determined by the sponsor according to the following criteria for each diagnosis:
  HAP/VAP/HCAP: Eradication was defined as the absence of the Baseline Gram-negative pathogen from an appropriate clinical specimen. If it was not possible to obtain an appropriate clinical culture and the participant had a successful clinical outcome, the response was presumed to be eradication.
  BSI/Sepsis: Absence of the Baseline Gram-negative pathogen from a blood culture and/or other primary source as applicable. In the case of sepsis, if the participant had a successful clinical outcome and it was not possible to obtain an appropriate clinical culture, the response was presumed to be eradication.
  cUTI: a urine culture that showed that the Gram-negative uropathogen identified at Baseline at ≥ 10⁵ CFU/mL was reduced to < 10³ CFU/mL.
  Overall per-participant eradication was defined as eradication of all Baseline Gram-negative pathogens.
Time Frame: End of treatment, Day 7 to 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 63 | 33 | 80 | 38
percentage of participants | 41.3 [29.0 to 54.4] | 27.3 [13.3 to 45.5] | 47.5 [36.2 to 59.0] | 26.3 [13.4 to 43.1]

23. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at TOC in Participants With HAP/VAP/HCAP + BSI/Sepsis, and Overall
Description: as for outcome 22
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 63 | 33 | 80 | 38
percentage of participants | 25.4 [15.3 to 37.9] | 24.2 [11.1 to 42.3] | 31.3 [21.3 to 42.6] | 23.7 [11.4 to 40.2]

24. Secondary Outcome: Percentage of Participants With Sustained Microbiologic Eradication at Follow-up in Participants With HAP/VAP/HCAP + BSI/Sepsis, and Overall
Description: Microbiological outcomes per Baseline pathogen at FU were determined according to the following criteria for each diagnosis:
  HAP/VAP/HCAP: Sustained eradication was defined as the absence of the Baseline Gram-negative pathogen from an appropriate clinical specimen after TOC.
  BSI/Sepsis: Absence of the Baseline Gram-negative pathogen from a blood culture or other primary source after TOC as applicable.
  For HAP/VAP/HCAP and sepsis if an appropriate clinical culture could not be obtained and the participant had a successful clinical response after TOC, the response was presumed sustained eradication.
  cUTI: a culture taken any time after documented eradication at TOC, and a urine culture obtained at FU showed that the Baseline uropathogen found at entry at ≥10⁵ CFU/mL remained < 10³ CFU/mL.
  Overall per-participant response was defined as sustained eradication of all Baseline Gram-negative pathogens after documented eradication at TOC.
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 63 | 33 | 80 | 38
percentage of participants | 22.2 [12.7 to 34.5] | 18.2 [7.0 to 35.5] | 26.3 [17.0 to 37.3] | 18.4 [7.7 to 34.3]

25. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at EOT By Baseline Pathogen
Description: as for outcome 22
Time Frame: End of treatment, Day 7 to 14
Population: Carbapenem-resistant Microbiological Intent-to-treat Population with the relevant Gram-negative pathogen at Baseline; participants with missing data were considered non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 34.6 | 30.0 | 60.0 | 28.6 | 0.0 |  | 41.7 | 29.4 | 40.5 | 29.4
  Pseudomonas aeruginosa: number analyzed (Participants) | 11 | 6 | 2 | 3 | 4 | 2 | 13 | 9 | 17 | 11
  Pseudomonas aeruginosa | 36.4 | 33.3 | 0.0 | 33.3 | 50.0 | 50.0 | 30.8 | 33.3 | 35.3 | 36.4
  Klebsiella pneumoniae: number analyzed (Participants) | 10 | 5 | 11 | 4 | 11 | 3 | 21 | 9 | 32 | 12
  Klebsiella pneumoniae | 50.0 | 20.0 | 72.7 | 25.0 | 81.8 | 0.0 | 61.9 | 22.2 | 68.8 | 16.7
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 20.0 |  |  |  |  |  | 20.0 |  | 20.0 |
  Escherichia coli: number analyzed (Participants) | 2 | 2 | 2 | 0 | 1 | 0 | 4 | 2 | 5 | 2
  Escherichia coli | 100.0 | 0.0 | 100.0 |  | 100.0 |  | 100.0 | 0.0 | 100.0 | 0.0

26. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at TOC By Baseline Pathogen
Description: as for outcome 22
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 30.8 | 30.0 | 20.0 | 28.6 | 0.0 |  | 27.8 | 29.4 | 27.0 | 29.4
  Pseudomonas aeruginosa: number analyzed (Participants) | 11 | 6 | 2 | 3 | 4 | 2 | 13 | 9 | 17 | 11
  Pseudomonas aeruginosa | 9.1 | 16.7 | 0.0 | 0.0 | 25.0 | 50.0 | 7.7 | 11.1 | 11.8 | 18.2
  Klebsiella pneumoniae: number analyzed (Participants) | 10 | 5 | 11 | 4 | 11 | 3 | 21 | 9 | 32 | 12
  Klebsiella pneumoniae | 50.0 | 20.0 | 54.5 | 50.0 | 72.7 | 0.0 | 38.1 | 33.3 | 50.0 | 25.0
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 0.0 |  |  |  |  |  | 0.0 |  | 0.0 |
  Escherichia coli: number analyzed (Participants) | 2 | 2 | 2 | 0 | 1 | 0 | 4 | 2 | 5 | 2
  Escherichia coli | 50.0 | 0.0 | 100.0 |  | 0.0 |  | 50.0 | 0.0 | 40.0 | 0.0

27. Secondary Outcome: Percentage of Participants With Sustained Microbiologic Eradication at Follow-up By Baseline Pathogen
Description: as for outcome 24
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 25
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 26.9 | 20.0 | 20.0 | 14.3 | 0.0 |  | 25.0 | 17.6 | 24.3 | 17.6
  Pseudomonas aeruginosa: number analyzed (Participants) | 11 | 6 | 2 | 3 | 4 | 2 | 13 | 9 | 17 | 11
  Pseudomonas aeruginosa | 9.1 | 16.7 | 0.0 | 0.0 | 0.0 | 50.0 | 7.7 | 11.1 | 5.9 | 18.2
  Klebsiella pneumoniae: number analyzed (Participants) | 10 | 5 | 11 | 4 | 11 | 3 | 21 | 9 | 32 | 12
  Klebsiella pneumoniae | 20.0 | 20.0 | 45.5 | 50.0 | 63.6 | 0.0 | 33.3 | 33.3 | 43.8 | 25.0
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 0.0 |  |  |  |  |  | 0.0 |  | 0.0 |
  Escherichia coli: number analyzed (Participants) | 2 | 2 | 2 | 0 | 1 | 0 | 4 | 2 | 5 | 2
  Escherichia coli | 50.0 | 0.0 | 50.0 |  | 0.0 |  | 50.0 | 0.0 | 40.0 | 0.0

28. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at EOT By Baseline Carbapenem-resistant Pathogen
Description: Microbiological outcome per Baseline carbapenem-resistant pathogen were determined according to the following criteria for each diagnosis:
  HAP/VAP/HCAP: Eradication was defined as the absence of the Baseline Gram-negative pathogen from an appropriate clinical specimen. If it was not possible to obtain an appropriate clinical culture and the participant had a successful clinical outcome, the response was presumed to be eradication.
  BSI/Sepsis: Absence of the Baseline Gram-negative pathogen from a blood culture and/or other primary source as applicable. In the case of sepsis, if the participant had a successful clinical outcome and it was not possible to obtain an appropriate clinical culture, the response was presumed to be eradication.
  cUTI: a urine culture that showed that the Gram-negative uropathogen identified at Baseline at ≥ 10⁵ CFU/mL was reduced to < 10³ CFU/mL.
  Overall per-participant eradication was defined as eradication of all Baseline Gram-negative pathogens.
Time Frame: End of treatment, Day 7 to 14
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 34.6 | 30.0 | 60.0 | 28.6 | 0.0 |  | 41.7 | 29.4 | 40.5 | 29.4
  Klebsiella pneumoniae: number analyzed (Participants) | 6 | 5 | 10 | 4 | 11 | 3 | 16 | 9 | 27 | 12
  Klebsiella pneumoniae | 33.3 | 20.0 | 70.0 | 75.0 | 81.8 | 0.0 | 56.3 | 22.2 | 66.7 | 16.7
  Pseudomonas aeruginosa: number analyzed (Participants) | 6 | 5 | 2 | 3 | 4 | 2 | 8 | 8 | 12 | 10
  Pseudomonas aeruginosa | 33.3 | 40.0 | 0.0 | 33.3 | 50.0 | 50.0 | 25.0 | 37.5 | 33.3 | 40.0
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 20.0 |  |  |  |  |  | 20. |  | 20.0 |

29. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at TOC By Baseline Carbapenem-resistant Pathogen
Description: as for outcome 28
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 30.8 | 30.0 | 20.0 | 28.6 | 0.0 |  | 27.8 | 29.4 | 27.0 | 29.4
  Klebsiella pneumoniae: number analyzed (Participants) | 6 | 5 | 10 | 4 | 11 | 3 | 16 | 9 | 27 | 12
  Klebsiella pneumoniae | 0.0 | 20.0 | 50.0 | 50.0 | 72.7 | 0.0 | 31.3 | 33.3 | 48.1 | 25.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 6 | 5 | 2 | 3 | 4 | 2 | 8 | 8 | 12 | 10
  Pseudomonas aeruginosa | 0.0 | 20.0 | 0.0 | 0.0 | 25.0 | 50.0 | 0.0 | 12.5 | 8.3 | 20.0
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 0.0 |  |  |  |  |  | 0.0 |  | 0.0 |

30. Secondary Outcome: Percentage of Participants With Sustained Microbiologic Eradication at Follow-up By Baseline Carbapenem-resistant Pathogen
Description: as for outcome 24
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 14
Measure: Number; unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants
  Acinetobacter baumannii: number analyzed (Participants) | 26 | 10 | 10 | 7 | 1 | 0 | 36 | 17 | 37 | 17
  Acinetobacter baumannii | 26.9 | 20.0 | 20.0 | 14.3 | 0.0 |  | 25.0 | 17.6 | 24.3 | 17.6
  Klebsiella pneumoniae: number analyzed (Participants) | 6 | 5 | 10 | 4 | 11 | 3 | 16 | 9 | 27 | 12
  Klebsiella pneumoniae | 0.0 | 20.0 | 40.0 | 50.0 | 63.6 | 0.0 | 25.0 | 33.3 | 40.7 | 25.0
  Pseudomonas aeruginosa: number analyzed (Participants) | 6 | 5 | 2 | 3 | 4 | 2 | 8 | 8 | 12 | 10
  Pseudomonas aeruginosa | 0.0 | 20.0 | 0.0 | 0.0 | 0.0 | 50.0 | 0.0 | 12.5 | 0.0 | 20.0
  Stenotrophomonas maltophilia: number analyzed (Participants) | 5 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 5 | 0
  Stenotrophomonas maltophilia | 0.0 |  |  |  |  |  | 0.0 |  | 0.0 |

31. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at EOT in Participants With Documented Carbapenem-resistant Gram-negative Bacteremia
Description: The percentage of participants who experienced eradication of the Baseline documented carbapenem-resistant Gram-negative bacteremia, defined as absence of the Baseline Gram-negative pathogen from a blood culture.
Time Frame: End of treatment, Day 7 to 14
Population: Carbapenem-resistant Microbiological Intent-to-treat Population with documented carbapenem-resistant Gram-negative bacteremia at Baseline (all infection sites combined); participants with missing data were considered non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cefiderocol | Best Available Therapy (BAT)
Number analyzed (Participants) | 22 | 13
percentage of participants | 54.5 [32.2 to 75.6] | 30.8 [9.1 to 61.4]

32. Secondary Outcome: Percentage of Participants With Microbiologic Eradication at TOC in Participants With Documented Carbapenem-resistant Gram-negative Bacteremia
Description: as for outcome 31
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentge of participants
Arm/Group | Cefiderocol | Best Available Therapy (BAT)
Number analyzed (Participants) | 22 | 13
percentge of participants | 31.8 [13.9 to 54.9] | 30.8 [9.1 to 61.4]

33. Secondary Outcome: Percentage of Participants With Sustained Microbiologic Eradication at Follow-up in Participants With Documented Carbapenem-resistant Gram-negative Bacteremia
Description: The percentage of participants who experienced sustained eradication of the Baseline documented carbapenem-resistant Gram-negative bacteremia, defined as absence of the Baseline Gram-negative pathogen from a blood culture after TOC.
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 31
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cefiderocol | Best Available Therapy (BAT)
Number analyzed (Participants) | 22 | 13
percentage of participants | 27.3 [10.7 to 50.2] | 23.1 [5.0 to 53.8]

34. Secondary Outcome: Percentage of Participants With a Composite Clinical and Microbiological Response at EOT
Description: The composite clinical and microbiological response rate is defined as the percentage of participants with both clinical cure and microbiologic eradication, as defined above for each site of infection.
Time Frame: End of treatment, Day 7 to 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants | 30.0 [16.6 to 46.5] | 26.3 [9.1 to 51.2] | 56.5 [34.5 to 76.8] | 21.4 [4.7 to 50.8] | 70.6 [44.0 to 89.7] | 20.0 [0.5 to 71.6] | 39.7 [27.6 to 52.8] | 24.2 [11.1 to 42.3] | 46.3 [35.0 to 57.8] | 23.7 [11.4 to 40.2]

35. Secondary Outcome: Percentage of Participants With a Composite Clinical and Microbiological Response at TOC
Description: as for outcome 34
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants | 22.5 [10.8 to 38.5] | 21.1 [6.1 to 45.6] | 30.4 [13.2 to 52.9] | 21.4 [4.7 to 50.8] | 47.1 [23.0 to 72.2] | 20.0 [0.5 to 71.6] | 25.4 [15.3 to 37.9] | 21.2 [9.0 to 38.9] | 30.0 [20.3 to 41.3] | 21.1 [9.6 to 37.3]

36. Secondary Outcome: Percentage of Participants With a Composite Clinical and Microbiological Response at Follow-up
Description: The composite clinical and microbiological response rate is defined as the percentage of participants with both sustained clinical cure and sustained microbiologic eradication, as defined above for each site of infection.
Time Frame: Follow-up, defined as 14 days after the end of treatment, equivalent to Study Day 21 to 28
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 63 | 33 | 80 | 38
percentage of participants | 20.0 [9.1 to 35.6] | 15.8 [3.4 to 39.6] | 26.1 [10.2 to 48.4] | 14.3 [1.8 to 42.8] | 41.2 [18.4 to 67.1] | 20.0 [0.5 to 71.6] | 22.2 [12.7 to 34.5] | 15.2 [5.1 to 31.9] | 26.3 [17.0 to 37.3] | 15.8 [6.0 to 31.3]

37. Secondary Outcome: All-cause Mortality at Day 14 and Day 28
Description: The all-cause mortality rate at Day 14 and Day 28 was calculated as the percentage of participants who experienced mortality regardless of the cause at or before Day 14 and Day 28, respectively.
Time Frame: Day 14 and Day 28
Population: The safety population includes randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | HAP/VAP/HCAP + BSI/Sepsis: Cefiderocol | HAP/VAP/HCAP + BSI/Sepsis: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 45 | 22 | 30 | 17 | 26 | 10 | 75 | 39 | 101 | 49
percentage of participants
  Day 14 | 24.4 [12.9 to 39.5] | 13.6 [2.9 to 34.9] | 16.7 [5.6 to 34.7] | 5.9 [0.1 to 28.7] | 11.5 [2.4 to 30.2] | 20.0 [2.5 to 55.6] | 21.3 [12.7 to 32.3] | 10.3 [2.9 to 24.2] | 18.8 [11.7 to 27.8] | 12.2 [4.6 to 24.8]
  Day 28 | 31.1 [18.2 to 46.6] | 18.2 [5.2 to 40.3] | 23.3 [9.9 to 42.3] | 17.6 [3.8 to 43.4] | 15.4 [4.4 to 34.9] | 20.0 [2.5 to 55.6] | 28.0 [18.2 to 39.6] | 17.9 [7.5 to 33.5] | 24.8 [16.7 to 34.3] | 18.4 [8.8 to 32.0]

38. Secondary Outcome: Percentage of Participants Alive and With No Change in Antibiotic Treatment Due to Either Lack of Therapeutic Benefit or Drug-related Toxicity at TOC
Time Frame: Test of cure, defined as 7 days after end of treatment, equivalent to Study Day 14 to 21
Population: Carbapenem-resistant Microbiological Intent-to-treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cefiderocol | Best Available Therapy (BAT)
Number analyzed (Participants) | 80 | 38
percentage of participants | 62.5 [51.0 to 73.1] | 60.5 [43.4 to 76.0]

39. Secondary Outcome: Survival Time
Description: Survival time was analyzed by Kaplan-Meier survival curve. The table below presents deaths that occurred in10-day time intervals through the end of study
Time Frame: Days 1 to 10, 11 to 20, 21 to 30, 31 to 40, 41-50, and 51 to 60.
Population: Carbapenem-resistant Microbiological Intent-to-treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | Cefiderocol | Best Available Therapy (BAT)
Number analyzed (Participants) | 80 | 38
Participants
  Days 1 to 10 | 12 | 3
  Days 11 to 20 | 9 | 3
  Days 21 to 30 | 1 | 2
  Days 31 to 40 | 4 | 0
  Days 41 to 50 | 1 | 0
  Days 51 to 60 | 0 | 0

40. Secondary Outcome: Change From Baseline in Clinical Pulmonary Infection Score (CPIS) in Participants With Pneumonia (HAP/VAP/HCAP)
Description: Clinical pulmonary infection score (CPIS) is a surrogate for diagnosis and treatment response. Points (0, 1, or 2) are assigned for observed findings for 5 variables including body temperature, white blood cell count, tracheal secretions, ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2), and chest radiograph infiltrates. The total score ranges from 0 to 10, where higher scores may indicate a higher likelihood of mortality; a negative change from Baseline indicates improvement
Time Frame: Baseline, end of treatment (Day 7-14), test of cure (7 days after end of treatment, equivalent to Study Day 14 to 21) and follow-up (14 days after end of treatment, equivalent to Study Day 21 to 28)
Population: Carbapenem-resistant microbiological intention-to-treat population; Participants with pneumonia and CPIS measurement at Baseline and at each post-baseline time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy
Number analyzed (Participants) | 39 | 18
scores on a scale
  End of treatment: number analyzed (Participants) | 33 | 17
  End of treatment | -2.5 (2.2) | -1.9 (1.7)
  Test of cure: number analyzed (Participants) | 27 | 14
  Test of cure | -3.1 (2.1) | -2.7 (2.2)
  Follow-up: number analyzed (Participants) | 26 | 13
  Follow-up | -3.4 (1.8) | -2.7 (1.9)

41. Secondary Outcome: Change From Baseline in Sequential Organ Failure Assessment (SOFA)
Description: The SOFA score is a scoring system to determine the extent of a patient's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal, and neurological systems. Each score is from 0 to 4, and the total score ranges from 0 to 24, where higher scores indicate a higher likelihood of mortality. A negative change from Baseline score indicates improvement.
Time Frame: Baseline, end of treatment (Day 7 to 14), test of cure (7 days after end of treatment, equivalent to Study Day 14 to 21) and follow-up (14 days after end of treatment, equivalent to Study Day 21 to 28)
Population: Carbapenem-resistant microbiological intention-to-treat population with SOFA measurement at Baseline and at each post-baseline time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | HAP/VAP/HCAP: Cefiderocol | HAP/VAP/HCAP: Best Available Therapy | BSI/Sepsis: Cefiderocol | BSI/Sepsis: Best Available Therapy | cUTI: Cefiderocol | cUTI: Best Available Therapy | Overall: Cefiderocol | Overall: Best Available Therapy
Number analyzed (Participants) | 40 | 19 | 23 | 14 | 17 | 5 | 80 | 38
scores on a scale
  End of treatment: number analyzed (Participants) | 33 | 18 | 19 | 14 | 14 | 3 | 66 | 35
  End of treatment | -0.7 (3.6) | -1.6 (2.6) | -2.1 (3.7) | -0.2 (2.8) | -0.6 (1.3) | -1.3 (2.3) | -1.1 (3.3) | -1.0 (2.7)
  Test of cure: number analyzed (Participants) | 27 | 14 | 14 | 11 | 15 | 3 | 56 | 28
  Test of cure | -1.3 (5.0) | -1.7 (2.9) | -2.1 (2.5) | 0.2 (4.1) | -0.6 (2.0) | -1.3 (2.3) | -1.3 (3.8) | -0.9 (3.4)
  Follow-up: number analyzed (Participants) | 26 | 14 | 15 | 9 | 13 | 3 | 54 | 26
  Follow-up | -2.1 (4.4) | -2.0 (2.9) | -3.1 (3.1) | -0.2 (4.4) | -0.1 (2.5) | -2.0 (3.5) | -1.9 (3.8) | -1.4 (3.5)

42. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity of each adverse event (AE) was graded by the investigator according to the following definitions:
  * Mild: Symptom or finding is minor and does not interfere with usual daily activities
  * Moderate: The event causes discomfort and interferes with usual daily activity or affects clinical status
  * Severe: The event causes interruption of usual daily activities or has a clinically significant effect
  The relationship of AEs to study treatment was determined by the investigator according to the following definition:
  ● Related: An AE which can be reasonably explained as having been caused by the study treatment.
  A serious AE is defined as any AE that resulted in any of the following outcomes:
  * Death
  * Life-threatening condition
  * Hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability/incapacity
  * Congenital anomaly/birth defect
  * Other medically important condition
Time Frame: From first dose of study drug up to 28 days after last dose; maximum treatment duration was 29 days in the cefiderocol group and 22 days in the BAT group.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Cefiderocol | Best Available Therapy (BAT)
Number analyzed (Participants) | 101 | 49
Participants
  Any adverse event (AE) | 92 | 47
  Mild adverse events | 23 | 9
  Moderate adverse events | 26 | 16
  Severe adverse events | 43 | 22
  Drug-related adverse events | 15 | 11
  Discontinuations due to adverse events | 10 | 3
  Discontinuations due to drug-related AEs | 3 | 2
  Serious adverse events (SAE) | 50 | 23
  Drug-related serious adverse events | 1 | 5
  Death due to serious adverse events | 34 | 9

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 days after last dose; For patients with HAP/VAP/HCAP or BSI/sepsis median treatment duration was 11.0 (2-22) days (cefiderocol) and 13.0 (2-22) days (BAT); In patients with cUTI median treatment duration was 10.5 (2-29) days (cefiderocol) and 6.5 (2-14) days (BAT).
Arm/Group | Cefiderocol | Best Available Therapy (BAT)
All-Cause Mortality (participants affected / at risk) | 34/101 | 9/49
Serious Adverse Events (participants affected / at risk) | 50/101 | 23/49
Other Adverse Events (participants affected / at risk) | 88/101 | 43/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cefiderocol (N=101) | Best Available Therapy (BAT) (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac arrest (Cardiac disorders) | 4 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 2 | 2
Pyrexia (General disorders) | 3 | 0
Sudden death (General disorders) | 1 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 3 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 2 | 0
Meningitis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Osteomyelitis acute (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Renal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 12 | 6
Systemic candida (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Liver function test abnormal (Investigations) | 4 | 3
Transaminases increased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 2 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Quadriplegia (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 2
Anuria (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 1
Shock (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cefiderocol (N=101) | Best Available Therapy (BAT) (N=49)
Anaemia (Blood and lymphatic system disorders) | 8 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 1
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 4
Thrombocytosis (Blood and lymphatic system disorders) | 3 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 3 | 2
Cyanosis (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 2
Hypothyroidism (Endocrine disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 1
Pupils unequal (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 8 | 3
Diarrhoea (Gastrointestinal disorders) | 19 | 6
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 7 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 13 | 7
Asthenia (General disorders) | 2 | 1
Catheter site inflammation (General disorders) | 0 | 1
Chest pain (General disorders) | 6 | 0
Fatigue (General disorders) | 1 | 2
Hypothermia (General disorders) | 2 | 1
Localised oedema (General disorders) | 1 | 1
Malaise (General disorders) | 1 | 1
Oedema (General disorders) | 4 | 0
Oedema peripheral (General disorders) | 5 | 2
Pain (General disorders) | 2 | 1
Pyrexia (General disorders) | 12 | 6
Biliary dilatation (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 1
Gallbladder necrosis (Hepatobiliary disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 0 | 1
Acinetobacter infection (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial disease carrier (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 3 | 0
Candida infection (Infections and infestations) | 4 | 1
Candiduria (Infections and infestations) | 2 | 1
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 2 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Corynebacterium infection (Infections and infestations) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Enterobacter infection (Infections and infestations) | 0 | 1
Enterococcal infection (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 2 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 2 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 1
Pseudomonas infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 3
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 3 | 1
Tracheobronchitis (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 2
Urinary tract infection enterococcal (Infections and infestations) | 3 | 0
Wound infection pseudomonas (Infections and infestations) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 4 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 7 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 1
Blood bilirubin increased (Investigations) | 2 | 1
Blood creatine increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 4 | 2
Blood lactate dehydrogenase increased (Investigations) | 1 | 1
Blood lactic acid increased (Investigations) | 1 | 1
Blood magnesium decreased (Investigations) | 3 | 0
Blood phosphorus decreased (Investigations) | 0 | 2
Blood urea increased (Investigations) | 1 | 1
Gastrointestinal stoma output increased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 2 | 1
Lipase increased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 4 | 1
Platelet count decreased (Investigations) | 0 | 2
White blood cell count abnormal (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 2
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 6
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 2 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 2
Metabolic alkalosis (Metabolism and nutrition disorders) | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2
Dizziness postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1
Agitation (Psychiatric disorders) | 5 | 2
Anxiety (Psychiatric disorders) | 2 | 2
Confusional state (Psychiatric disorders) | 2 | 1
Delirium (Psychiatric disorders) | 4 | 0
Depression (Psychiatric disorders) | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 3
Restlessness (Psychiatric disorders) | 3 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 4
Bladder disorder (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 2 | 2
Renal disorder (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Genital erythema (Reproductive system and breast disorders) | 0 | 1
Oedema genital (Reproductive system and breast disorders) | 0 | 1
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 10 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 4
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 6 | 2
Shock (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can embargo results from a PI's center until the combined results from the completed study have been published in full or the sponsor confirms there will be no multicenter study publication. Results communications must be provided to the sponsor for review at least 60 days before submission for publication. By written request, the sponsor can extend the embargo up to an additional 60 days. The sponsor cannot require changes to scientific content and cannot further extend the embargo.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-27): https://cdn.clinicaltrials.gov/large-docs/95/NCT02714595/SAP_000.pdf
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT02714595/Prot_001.pdf